CLINICAL TRIAL: NCT01048684
Title: Comparison of Two Doses of Mannitol on Brain Relaxation During Supratentorial Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: François Girard MD FRCPC, Centre de recherche du CHUM (CRCHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG2010-003
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Brain Tumor; Intracranial Pressure
Keywords: Brain tumor; Intracranial pressure
MeSH Terms: conditions — Brain Neoplasms | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20% Mannitol 0.7 g/kg (low-dose) (Active Comparator): Study subjects will be randomized to receive an infusion of 20% mannitol 0.7g/kg over 30 minutes after induction of general anesthesia.
  Interventions: Drug: Mannitol
- 20% Mannitol 1.4 g/kg (high dose) (Experimental): Study subjects will be randomized to receive an infusion of 20% mannitol 1.4 g/kg over 30 minutes after induction of general anesthesia.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — Variation of mannitol dose
  Arms: 20% Mannitol 0.7 g/kg (low-dose)
Drug: Mannitol — Variation of mannitol dose
  Arms: 20% Mannitol 1.4 g/kg (high dose)

SUMMARY:
Neuroanesthesia for supratentorial surgery involves a thorough understanding of the physiopathology of intracranial pressure, cerebral homeostasis and regulation of cerebral perfusion pressure as well as the effects of anesthesia and surgery on these elements.

The main objective of anesthesia during neurosurgery is to preserve the integrity of the brain by maintaining cerebral homeostasis, and assuring cerebral protection using normovolemia, normotension, normoglycemia, moderate hyperoxia and hypocapnia and hyperosmolality with the administration of mannitol.

During surgery, the use of surgical retractors must be limited to avoid possible ischemia of the brain tissue. Surgical retractors can be replaced by chemical retractors. The concept of chemical retraction involves a reduction of cerebral blood flow, maintaining cerebral perfusion pressure, moderate hyperventilation, drainage of cerebrospinal fluid and osmotherapy.

Mannitol, an osmotic agent, has been widely used to reduce the volume of the brain, the intracranial pressure and to facilitate the surgical approach in reducing the risk of cortical lesions during the opening of the skull.

Mannitol 20% is usually given intravenously in bolus doses of 0.5-1g/kg over 30 minutes. However, over the last few years, the concept of a dose-response relationship has emerged. Some recent studies tend to demonstrate that higher doses of mannitol could reduce intracranial pressure significantly without any important side effects.

The main objective of the present study is to compare two doses of mannitol (0.7 and 1.4 g/kg) on brain relaxation during supratentorial craniotomies.

DETAILED DESCRIPTION:
80 patients will be divided in two equal groups (Group 1: to receive 20% mannitol 0.7 g/kg or Group 2: 1.4 g/kg).

The anesthetic technique and monitoring will be standardized. The administration of mannitol will start following the induction of general anesthesia. The infusion will be given intravenously over 30 minutes.

Brain relaxation will be assessed by a senior surgeon at the opening of the dura mater on a scale from 1 to 4 (1= perfectly relaxed, 2= satisfactorily relaxed, 3= firm brain, 4=bulging brain)

If needed, in case of significant cerebral edema, a rescue dose of 20% mannitol 0.25 g/kg will be administered.

Hemodynamic variables (MAP, heart rate), temperature, urine output, perioperative fluid balance, blood loss and laboratory values (blood gases, electrolytes, osmolality, hematocrit, glycemia, lactates) will be collected immediately prior to the infusion of mannitol and at 30, 60, 180 minutes following the administration of mannitol.

The type of cerebral lesion, its location and size (in 3 dimensions) will be noted. The presence of a median-line shift will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patients who are to undergo an elective supratentorial craniotomy
* Physical status ASA I to IV inclusive.

Exclusion Criteria:

* Pregnancy
* Severe congestive heart failure
* Severe chronic renal failure
* Recent use (less than 24 hours before surgery)of mannitol or other hypertonic solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Brain relaxation at the opening of the dura mater assessed by a senior surgeon on a scale from 1 to 4 (1= perfectly relaxed, 2= satisfactorily relaxed, 3= firm brain, 4=bulging brain) | At the opening of the dura mater

SECONDARY OUTCOMES:
Hemodynamic variables: MAP, heart rate | Immediately prior to the infusion of mannitol and at 30, 60, 180 minutes after the administration of mannitol
Temperature | Immediately prior to the infusion of mannitol and at 30, 60, 180 minutes after the administration of mannitol
Urine output | Immediately prior to the infusion of mannitol and at 30, 60, 180 minutes after the administration of mannitol
Perioperative fluid balance and blood loss | Immediately prior to the infusion of mannitol and at 30, 60, 180 minutes after the administration of mannitol
Laboratory data: blood gases, electrolytes, osmolality, hematocrit, glycemia, lactates | Immediately prior to the infusion of mannitol and at 30, 60, 180 minutes after the administration of mannitol

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada